CLINICAL TRIAL: NCT06425380
Title: Pilot Open-Label Trial of Resistant Potato Starch in Patients With Cirrhosis and Overt Hepatic Encephalopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patricia P. Bloom, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-005555
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: Resistant Potato Starch
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resistant potato starch (Experimental): This will be taken for four weeks by enrolled participants.
  Interventions: Other: Resistant Potato Starch

INTERVENTIONS:
Other: Resistant Potato Starch — Participants will receive 4 weeks of resistant potato starch 20 grams (g) twice daily. Bob's Red Mill® potato starch will be used. Every patient will receive the same dose and there are no dose titrations.

SUMMARY:
This research is studying how a food product (resistant potato starch) which is a dietary supplement made from potato starch affects the gut bacteria of people with cirrhosis and hepatic encephalopathy.

The researchers in this study want to understand how potato starch works in the subject's body and how the body will react to it. Along with taking the study product participants health-related information and stool will be collected for this research study.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent, with signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Diagnosis of cirrhosis based on liver biopsy, imaging, or evidence of clinical decompensation.
* History of at least one episode of overt Hepatic Encephalopathy (HE) in the last year.

  * Defined by West Haven Criteria Grades II to IV
  * Can be precipitated Hepatic Encephalopathy (HE) episode.
* Sexually active women of childbearing potential enrolled in the study must agree to use a highly-effective method of contraception (defined in the protocol) for the duration of the study.

Exclusion Criteria:

* Hospitalization in the last 4 weeks
* Current refractory ascites (requiring large volume paracentesis to manage ascites)
* Gut-absorbable or intravenous antibiotic therapy in the last 4 weeks (rifaximin is permitted)
* Anticipated antibiotics in the coming 4 weeks
* Use of lactulose in the last 4 weeks
* Alcohol or illicit drug intake in the last 4 weeks

  * By history
  * Alcohol use will be characterized as >1 alcoholic drink / week
* History of inflammatory bowel disease
* History of primary sclerosing cholangitis
* Total bilirubin in the last 3 months > 4 mg/dL
* Prior diagnosis of dementia or other primary neurocognitive disorder
* Pregnancy or breast feeding
* Placement of a portosystemic shunt or transjugular intrahepatic portosystemic shunt in the last 3 months (permissible if placed >3 months before enrollment)
* Allergy to resistant potato starch

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in stool short-chain fatty acid (SCFA) levels from baseline to week 4 | Baseline, Week 4
  The study team will compare the total concentrations of the 3 most abundant SCFAs in humans (acetate, propionate, and butyrate) at baseline and week 4. Stool will undergo SCFA quantification by the University of Michigan Metabolomics core.

SECONDARY OUTCOMES:
Change in animal naming test (ANT) from baseline to week 4 | Baseline, Week 4
  In this test patients name as many animals as they can in 60 seconds. The ANT score is the number of unique animals named.
Number and type of adverse events from baseline to week 8 | baseline to week 8
  The severity or grade of an adverse event may be measured using the following definitions:
  Mild: Noticeable to the subject, but does not interfere with subject's expected daily activities, usually does not require additional therapy or intervention, dose reduction, or discontinuation of the study.
  Moderate: Interferes with the subject's expected daily activities, may require some additional therapy or intervention but does not require discontinuation of the study.
  Severe: Extremely limits to the subject's daily activities and may require discontinuation of study therapy, and/or additional treatment or intervention to resolve and may be life-threatening or fatal.
Change in T-score for the Patient Reported Outcomes Measurement Information System (PROMIS) gastrointestinal diarrhea 6a baseline to week 4 | Baseline, Week 4
  Gastrointestinal questionnaire has six questions with a total score ranging from 1-30 with the lower score indicating a healthier status.
Change in T-score for the PROMIS Gastrointestinal Gas and Bloating 13a scale baseline to week 4 | Baseline, Week 4
  The Gas and Bloating scale has13 questions (scale 2-60; with higher scores corresponding to more severe gas/bloating).
Number of patients enrolled in the study as a proportion of the number of patients contacted by the study team | start of screening, end of enrollment (approximately 20 months)
Feasibility of completing study activities | baseline, week 8
  Proportion of study activities completed
Feasibility based on the number of specimens collected | baseline, week 4
  Proportion of study samples collected (number collected from all patients / number requested from patients).
Retention to end of study | start of screening, end of enrollment (approximately 20 months)
  Proportion of drop outs
Intervention adherence | baseline, week 4
  Proportion of doses consumed

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bloom, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No